CLINICAL TRIAL: NCT00084734
Title: A Phase I and Pharmacokinetics Study of Docetaxel in Combination With Capecitabine and Cisplatin in Solid Tumors
Brief Title: Docetaxel, Capecitabine, and Cisplatin in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000365571; RPCI-RPC-0209
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Capecitabine; Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine — Oral
Drug: cisplatin — IV
Drug: docetaxel — IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, capecitabine, and cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one chemotherapy drug may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of docetaxel, capecitabine, and cisplatin in treating patients with metastatic or unresectable solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of docetaxel, cisplatin, and capecitabine in patients with advanced solid tumors.
* Determine the dose-limiting toxicity and recommended phase II dose of this regimen in these patients.

Secondary

* Determine the non-dose-limiting toxic effects associated with this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine any clinical activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive docetaxel IV over 30 minutes and cisplatin IV over 30 minutes on days 1 and 8 and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of docetaxel, cisplatin, and capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients receive treatment at the MTD.

PROJECTED ACCRUAL: A minimum of 21 patients will be accrued for this study within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor for which standard curative or palliative measures do not exist or are no longer effective

  * Metastatic or unresectable disease
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL

Hepatic

* AST and ALT ≤ 2.0 times upper limit of normal (ULN) AND alkaline phosphatase [AP] < ULN OR
* AP ≤ 4 times ULN AND AST and ALT < ULN
* Bilirubin normal

Renal

* Creatinine ≤ 1.5 mg/dL OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to ingest oral medications
* No allergy attributed to study drugs, compounds of similar chemical or biological composition, drugs formulated in polysorbate 80, or other agents used in this study
* No inner ear auditory toxicity ≥ grade 2
* No peripheral neuropathy ≥ grade 2
* No immunodeficiency
* No active or ongoing infection
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent growth factors (sargramostim [GM-CSF] or filgrastim [G-CSF])

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy and recovered

Surgery

* Not specified

Other

* No other concurrent investigational agents unless approved by the principal investigator and medical monitor
* No other concurrent anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2002-05; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of docetaxel, cisplatin, and capecitabine in patients with advanced solid tumors. | Every 21 days

SECONDARY OUTCOMES:
Determine the non-dose-limiting toxic effects associated with this regimen in these patients | Every 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States